CLINICAL TRIAL: NCT06810453
Title: The Effects of End-tidal Controlled Low-Flow Anesthesia on Anesthetic Agent Consumption in Elective Surgeries
Brief Title: The Effects of Sevoflurane and Desflurane Used in Low-Flow Anesthesia on Thiol Disulfide Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Elzem SEN, Assoc. Prof., University of Gaziantep
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020/283
Record Dates: First submitted 2025-01-14; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Low Flow Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane (Other): sevoflurane low-flow anesthesia
  Interventions: Other: A 5 cc venous blood sample was obtained; Procedure: low-flow anesthesia
- desflurane (Other): desflurane low-flow anesthesia
  Interventions: Other: A 5 cc venous blood sample was obtained; Procedure: low-flow anesthesia

INTERVENTIONS:
Other: A 5 cc venous blood sample was obtained — A 5 cc venous blood sample was obtained just before anesthesia induction and at the end of surgery.
Procedure: low-flow anesthesia — Low-flow anesthesia, also known as inhalational anesthesia method, is a type of anesthesia that is performed using a semi-closed, rebreathing system containing at least 50% fresh gas. Generally, low-flow anesthesia is used in anesthesia practices because it reduces costs, prevents environmental pollution, increases the humidity of gases, and reduces heat loss. Another important benefit of low-flow is that it requires closer monitoring of patients, which allows for early detection of complications during general anesthesia, thus improving patient safety. Concerns about low-flow anesthesia being used infrequently in the past have been addressed by the introduction of modern anesthesia workstations with sophisticated monitoring and safety features, which have made low-flow anesthesia widely used in most centers.

SUMMARY:
This study aimed to compare the effects of sevoflurane and desflurane used in low-flow anesthesia on thiol-disulfide homeostasis of patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Fifty patients were included who were scheduled to undergo elective total thyroidectomy operation under general anesthesia. The patients were assigned to one of 2 groups. Group S was the low-flow sevoflurane anesthesia group and Group D was the low-flow desflurane group. Blood samples were collected to evaluate thiol disulfide homeostasis preoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled to undergo elective total thyroidectomy under general anesthesia

Exclusion Criteria:

* Patients with diabetes mellitus, alcohol or drug addiction, smoking habits, expected difficult intubation, morbid obesity, chronic obstructive pulmonary disease, cardiovascular disease and those in pregnancy or lactation period were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Serum thiol-disulfide homeostasis parameters measurement/ calculation | A 5 cc venous blood sample was obtained just before the anesthesia induction and at the end of surgery.
  Serum thiol-disulfide homeostasis parameters were evaluated using an automated method (3). Homeostasis parameters include disulfide, native thiol (NT) and total thiol (TT) levels, and disulfide/TT, NT/TT, and disulfide/NT ratios. TT and NT levels were measured in μmol/L on a Beckman Coulter AU480 analyzer using a commercial kits (Rel Assay Diagnostics, Türkiye). The amount of disulfide was calculated using the formula ((TT-NT) /2). Then, ratios were calculated as percentages

CONTACTS AND LOCATIONS:
Overall Officials: Elzem Sen, Assoc Prof, Principal Investigator — University of Gaziantep
Locations (1):
- Elzem Sen, Gaziantep, Sehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No